CLINICAL TRIAL: NCT04792996
Title: Investigating the Preventive Potential of Bilirubin
Brief Title: Preventive Potential of Bilirubin
Acronym: BILIHEALTH
Status: Completed | Type: Observational
Sponsor: University of Vienna (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Wagner Karl-Heinz, Professor of Human Nutrition, University of Vienna
Other Study IDs: UNIVIE-BILIHEALTH
Record Dates: First submitted 2021-03-03; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Mild Hyperbilirubinaemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gilbert´s Syndrome: Subjects with mild hyperbilirubinaemia and a plasma level of unconjugated bilirubin of 17.1 µmol.
  Interventions: Other: No intervention
- Control group: Healthy controls with lower plasma level of unconjugated bilirubin of 17.1 µmol, aen and gender matched.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. case - control design.

SUMMARY:
The prevalence of mild hyperbilirubinemia, also known as Gilbert´s Syndrome, is usually defined using an unconjugated bilirubin (UCB) blood concentration above 17.1 µmol/l. The prevalence of GS is remarkably common, affecting 5-10% (depending on ethnicity and gender) of the adult population.

The aim of this project is to investigate whether there is a difference in health related marker between 60 subjects with Gilbert´s Syndrome (mild hyperbilirubinaemia) and 60 age and gender matched control subjects.

ELIGIBILITY:
Inclusion Criteria:

In general

* Signed declaration of consent
* Age: 20-80 years
* Liver enzymes (AST, ALT, GGT) < 1.5x over norm values
* Non smoking
* Moderate physical activity
* Ability to communicate with the study team in the local language to understand the study procedure

Cases (GS):

* Total blood bilirubin > 1.2 mg/dl
* Unconjugated bilirubin > 1 mg/dl

Controls (non-GS):

* Total blood bilirubin ≤ 1.2 mg/dl
* Unconjugated bilirubin ≤ 1 mg/dl

Exclusion Criteria:

In general

* Age < 20 or > 80 years
* Cardiovascular diseases
* Liver diseases (including Hep B and C)
* Cholelithiasis
* Hemolysis
* Renal diseases
* Active tumors
* Diabetes mellitus
* Smoking
* Professional athletes
* Subjects with organ transplants
* Intake of antioxidants within the last 4 weeks
* Intake of liver influencing medication within the last 5 weeks

Cases (GS):

* Total blood bilirubin ≤ 1.2 mg/dl
* Unconjugated bilirubin ≤ 1 mg/dl

Controls (non-GS):

* Total blood bilirubin > 1.2 mg/dl
* Unconjugated bilirubin > 1 mg/dl

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 120 participants, 60 participants with mild hyperbilirubinaemia, 60 subjects without mild hyperbilirubinaemia, age and gender matching.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
The investigators will consider Lipid parameter | Baseline
  Compare plasma parameter of lipid metabolism (Cholesterol, LDL, HDL, Triglycerides, ..) between Gilbert´s Syndrome subjects and controls.

SECONDARY OUTCOMES:
The investigators will consider plasma parameter of glucose metabolism | Baseline
  Compare plasma parameter of glucose metabolism (plasma glucose (mg/dl), plasma insulin (µU/ml), C-peptide (ng/ml)) between Gilbert´s Syndrome subjects and controls.
The investigators will consider AMPK metabolic pathway | Baseline
  Compare parameter of the AMPK metabolic pathway (phosphorylated AMPK (rfU), phosphorylated Ppar-alpha (rfU), phosphorylated Ppar-gamma (rfU)) between Gilbert´s Syndrome subjects and controls.
The investigators will consider body composition | Baseline
  Compare parameter of the body composition (BMI (kg/m2), fat mass (%), waist circumference (cm), hip circumference (cm), abdominal circumference (cm)) between Gilbert´s Syndrome subjects and controls.
The investigators will consider heme catabolic pathway | Baseline
  Compare parameter of the heme catabolic pathway (expression of heme oxygenase (RQ), expression of Biliverdinreductase (RQ)) between Gilbert´s Syndrome subjects and controls.
The investigators will consider the metabolomic response | Baseline
  Compare the metabolomic pattern (ie all metabolites; analyzed using both nuclear magnetic resonance (NMR) and mass spectrometry (MS) techniques) between Gilbert´s Syndrome subjects and controls.
The investigators will consider the composition of gut-microbiota | Baseline
  Compare the composition of the gut microbiota (Gene sequencing of the 16S rRNA on the stool samples are performed to identify the microbes down to genus level as well as the microbial diversity and relative abundance) between Gilbert´s Syndrome subjects and controls.
The investigators will consider oxidative stress marker | Baseline
  Compare plasma concentrations of oxidative stress marker such as malondialdehyde or GSH/GSSG between Gilbert´s Syndrome subjects and controls.
The investigators will consider anabolic and catabolic hormones | Baseline
  Compare plasma concentrations of hormones (Glucagon (pg/ml), T3 (pg/ml), TSH(µM/ml),) between Gilbert´s Syndrome subjects and controls.
The investigators will consider telomere length | Baseline
  Compare telomere length between Gilbert´s Syndrome subjects and controls.
The investigators will consider RNA and DNA gene expression | Baseline
  Compare RNA and DNA gene expression between Gilbert´s Syndrome subjects and controls.
The investigators will consider the metabolomic response after a standard breakfast | Five blood samplings over 180 minutes.
  Compare the metabolomic pattern after a standard breakfast (ie all metabolites; analyzed using both nuclear magnetic resonance (NMR) and mass spectrometry (MS) techniques) between Gilbert´s Syndrome subjects and controls.

IPD SHARING:
Plan to Share IPD: No